CLINICAL TRIAL: NCT04424004
Title: MURDOCK Cabarrus County COVID-19 Prevalence and Immunity (C3PI) Study
Acronym: C3PI
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pro00105703
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing; COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nose Swabs and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MURDOCK Study Participants with valid email address: Randomized for testing: 1.A randomly selected subset of individuals who consent to participate (N~300-500), will be invited to participate in COVID-19 polymerase chain reaction (PCR) viral testing by at-home collection and return of self-administered nasal swabs. Saliva specimens may replace the nasal swab specimen.
  2. The same randomly selected subset of individuals who collect at-home samples for COVID-19 PCR testing (N~300-500), will also provide a blood sample for serologic testing for SARS-CoV-2 IgG antibodies.
  Interventions: Other: COVID-19 PCR and serology testing

INTERVENTIONS:
Other: COVID-19 PCR and serology testing — 1. PCR testing: participate will conduct at-home collection and return of self-administered nasal swabs for COVID-19 polymerase chain reaction (PCR) viral testing. Saliva specimens may replace the nasal swab specimen. Specimens will be collected at baseline and every 2 weeks in conjunction with questionnaire administration.
  2. Serology testing: The same randomized participants will also provide a blood sample for serologic testing for SARS-CoV-2 IgG antibodies. Specimens will be collected by routine venipuncture at the MURDOCK Study office in Kannapolis, NC.Specimens for serology will be collected at baseline approximately 1 month after the first questionnaire and 2 weeks after the first nasal swab collection and COVID-19 PCR testing. Specimens for serology will be collected at least bi-monthly and up to monthly thereafter through a total study duration of 6, and up to 12, months.
  Other Names: COVID-19 PCR testing; COVID-19 serology testing

SUMMARY:
The objectives of this research is to:

* Assess perceptions, concerns, and practices related to the COVID-19 pandemic and mitigation strategies using the MURDOCK Study Community Registry and Biorepository population as a measure of these features in Cabarrus County through a biweekly electronic survey.
* Estimate the prevalence and change in prevalence of COVID-19 infection based on responses to questionnaire items on symptoms and practices using a biweekly electronic survey.
* Among respondents to the baseline questionnaire, conduct at home mid-turbinate nasal swab collection for viral PCR testing for active COVID-19 infection as an estimate of the prevalence of active infection in Cabarrus County.
* Among respondents to the baseline questionnaire, conduct serologic testing for IgG antibodies to SARS-CoV-2 as an estimate of the prevalence of exposure and potential immunity to COVID-19.

DETAILED DESCRIPTION:
Method:

Questionnaire The investigators will use RedCap to introduce the study, obtain online informed consent, and administer an electronic questionnaire to MURDOCK Study participants currently residing in North Carolina who have a valid email address on file (N~7200). The question bank for the questionnaire is attached to the application. It includes demographics, education and employment, and questions about symptoms, contacts and exposures, the participant's household, behaviors, and practice of mitigation strategies. The opportunity to enroll and complete the baseline questionnaire will remain open for 1 month. Follow up surveys will be made available to consented participants on the same day for each week they are administered. The investigators anticipate a 20% response rate to the survey (N~1500). Recruitment materials, consent and questionnaires, materials related to return of results to participants, and verbal study communications will be available in both English and Spanish.

COVID-19 PCR testing A randomly selected subset of individuals who consent to participate (N~300-500 initially, with the potential to expand testing to more survey participants as additional funding becomes available), weighted to ensure representation by race/ethnicity, age, and sex, will be invited to participate in COVID-19 polymerase chain reaction (PCR) viral testing by at-home collection and return of self-administered nasal swabs. Saliva specimens may replace the nasal swab specimen. Specimens will be collected at baseline and every 2 weeks in conjunction with questionnaire administration. Participants will have the opportunity to opt out of participation in this component at the time of consent and enrollment. Those who do not opt out will be eligible for the random selection for COVID-19 testing. The investigators will provide specimen collection materials and instructions for collection, along with return shipping instructions to participants in pre-prepared kits. COVID-19 PCR testing will be conducted at the North Carolina State Laboratory of Public Health. This is a CLIA-certified laboratory. Samples for COVID-19 PCR testing will be identified only by a unique study identification number for each participant. Results of COVID-19 testing will be returned from the State Lab to the MURDOCK Study investigative team as results are available from testing (expected turnaround time ~4 days from receipt at State Lab) by secure transfer for incorporation into the RedCap study database.

COVID-19 serology testing The same randomly selected subset of individuals who collect at-home samples for COVID-19 PCR testing (N~300-500 initially, with the potential expand to more survey participants as additional resources become available), will also provide a blood sample for serologic testing for SARS-CoV-2 IgG antibodies. Specimens will be collected by routine venipuncture at the MURDOCK Study office in Kannapolis, NC and potentially 2-3 additional locations in Cabarrus County. Study visits for venipuncture will be deferred for 2 weeks in participants whose nasal swab PCR testing for COVID-19 is positive. Participants will be screened for COVID-19 symptoms at the time of scheduling the visit for venipuncture and at arrival for the visit. Participants who screen positive for COVID-19 symptoms will be referred for clinical COVID-19 testing and will have their initial serology testing deferred until a negative clinical test is documented or for 2 weeks if clinical testing is not performed.

Specimens for serology will be collected at baseline approximately 1 month after the first questionnaire and 2 weeks after the first nasal swab collection and COVID-19 PCR testing. Specimens for serology will be collected at least bi-monthly and up to monthly thereafter through a total study duration of 6, and up to 12, months. SARS-CoV-2 serologic testing for IgG antibodies will be conducted in the laboratory of Thomas Denny, MSc, MPhil in the Duke Human Vaccine Institute on the campus of Duke University Medical Center using a commercial IgG assay (Perkin-Elmer). Samples for serology will be identified only by a unique study identification number for each participant. Results of serological testing will be returned from the Denny laboratory to the MURDOCK Study investigative team at regular, prespecified intervals by secure transfer for incorporation into the RedCap study database. The Denny laboratory is CLIA-certified. Any residual serum after SARS-CoV-2 serologic testing will be frozen at -80°C and stored for future use in the Duke COVID-19 Biorepository (Pro00105316).

Return of Results to Participants:

The investigators will share aggregate results from questionnaires and testing with all participants and the public through multiple routes, including email, social media and the press and with the scientific community through presentations at scientific meetings and publications. The investigators will also provide regular reports on accruing study data to NCDHHS. Participants will not be identified individually in these aggregate reports. The investigators also will return the results of both COVID-19 PCR testing and serologic testing for SARS-CoV-2 antibodies to individual study participants. Individual return of results will follow the following principles:

COVID-19 test results. A standard template for return of negative COVID-19 test results will be IRB approved and used to notify participants of their results. If a participant tests positive for COVID-19, the participant will be contacted by phone by the study PI or a designate to convey the result. General recommendations for participants who test positive will be IRB approved. The investigators will also offer these participants a link through which they can consider participation in the Duke COVID Community Watch support program (Pro00105189). Positive COVID-19 test results will also be reported to the local/state health department.

SARS-CoV-2 serology results. An IRB approved standard template will be used to convey the results of SARS-CoV-2 serology to participants. Care will be taken to ensure that participants understand what information the results of their SARS-CoV-2 serology conveys (and does not convey) in order to avoid any risk of misinterpretation, particularly of positive results.

Selection of Subjects

List inclusion/exclusion criteria and how subjects will be identified. The MURDOCK NCDHHS COVID-19 Prevalence Study will examine COVID-19 prevalence and SARS-CoV-2 antibody prevalence in Cabarrus County, NC by leveraging the community-based cohort enrolled in the MURDOCK Study Community Registry and Biorepository (MURDOCK Study). The MURDOCK Study is an ongoing longitudinal health study operated by the Translational Population Health Research Center in the Duke Clinical & Translational Science Institute and approved by the Duke University Institutional Review Board (Duke IRB Pro00011196). The MURDOCK Study recruited 12,526 residents from 20 Zip Codes in the Cabarrus County/Kannapolis region, and currently follows 10,407 active participants. As part of the MURDOCK Study, all participants provided demographic, clinical, and behavioral data via an enrollment questionnaire, were geospatially mapped at the street address level, and consented to a yearly follow up questionnaire. They also provided consent to be contacted by MURDOCK Study staff up to four times per year to consider participation in future research opportunities. A recent protocol communication to the IRB was approved to allow additional contacts for high priority COVID-19 research studies (Pro00011196-SE-45.0). Our study population for this protocol will include approximately 7200 active MURDOCK Study participants who currently reside in North Carolina and have a valid email address on file. The active study participants who receive a recruitment email and consent to participate (estimated 20%) will have the opportunity to declare their interest in testing and from among those 300-500 will be randomly selected to participate in the testing. The anticipated number to enroll is set at 1,000 but may be adjusted up based on response rate.

ELIGIBILITY:
Inclusion Criteria:

* MURDOCK Study participants ( Pro00011196) currently residing in North Carolina who have a valid email address on file.

Exclusion Criteria:

* MURDOCK Study participants ( Pro00011196) currently not residing in North Carolina
* MURDOCK Study participants without a valid email address on file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALL active MURDOCK study participants who currently reside in North Carolina and have a valid email address. The demographics of the MURDOCK study cohort are representative of the population in Cabarrus County and North Carolina.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Estimate the prevalence of COVID-19 infection based on responses to questionnaire items on symptoms and practices using a biweekly electronic survey. | 6 months
  RedCap link will be sent to participants electronically and they will complete and submit the questionnaire.
Assess perceptions, concerns, and practices related to the COVID-19 pandemic and mitigation strategies | 6 months
  This will be accomplished using the MURDOCK Study Community Registry and Biorepository (Pro00011196) population as a measure of these features in Cabarrus County through a biweekly electronic survey
Estimate of the prevalence of active infection in Cabarrus County. | 6 months
  Among respondents to the baseline questionnaire, conduct bi-weekly at home anterior nares swab collection for viral PCR testing for active COVID-19 infection
Estimate of the prevalence of exposure and potential immunity to COVID-19. | 6 months
  Among respondents to the baseline questionnaire, conduct bimonthly serologic testing for IgG antibodies to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Newby, MD, Principal Investigator — Duke University
Locations (1):
- Duke CTSI Translational Population Health Office, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No